CLINICAL TRIAL: NCT04204863
Title: Status Epilepticus Population Study (STEPS)
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-00693; me19Sutter5
Record Dates: First submitted 2019-12-17; First posted 2019-12-19 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Epileptic Seizures
Keywords: Status epilepticus; Electroencephalogram
MeSH Terms: conditions — Seizures; Status Epilepticus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- SE patients
  Interventions: Other: collection of patient data

INTERVENTIONS:
Other: collection of patient data — Extract data from the digital medical records, the electroencephalographic and microbiologic database.

SUMMARY:
The aim of this observational multicenter cohort study is to gain a deeper understanding regarding the effects of treatment adaption based on information from outcome prediction models, risk stratification, as well as treatment monitoring, detection, prevention, and management of complications on course and outcome of adult patients with status epilepticus (SE).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (i.e., patients ≥18 years of age) with diagnosed SE between 2005 and 2023 who have been treated at the University Hospital of Basel or the Cantonal Hospital Aarau.

Exclusion Criteria:

* Patients younger than 18 years.
* Patients with repetitive epileptic seizures not qualifying for SE.
* Patients with documented refusal of the general consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (i.e., patients ≥18 years of age) with SE treated at the University Hospital Basel and the Cantonal Hospital Aarau.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2019-04-19 (Actual); Primary Completion 2050-12 (Estimated); Study Completion 2050-12 (Estimated)

PRIMARY OUTCOMES:
Demographics | between 01.01.2005 and 31.12.2023
  age, sex
Data from acute prehospital management by the emergency medical services (EMS) | between 01.01.2005 and 31.12.2023
  extracted from the treatment protocols of the EMS
Duration of ICU (intensive care unit) and hospital stay, and destination at discharge | between 01.01.2005 and 31.12.2023
  Duration of ICU (intensive care unit) and hospital stay, and destination at discharge
Date(s) of seizure(s) captured by electroencephalographic (EEG) data | between 01.01.2005 and 31.12.2023
  Date(s) of seizure(s) captured by EEG
Seizure history and etiology | between 01.01.2005 and 31.12.2023
  withdrawal from anti seizure drugs, structural, infectious, or autoimmune causes
Number and Duration of SE episodes | between 01.01.2005 and 31.12.2023
  Number and Duration (time) of SE episodes
Types of SE | between 01.01.2005 and 31.12.2023
  Types of SE according to the current guidelines from the International League of Epilepsy (ILAE) (i.e., nonconvulsive with coma, SE with motor symptoms, focal nonconvulsive SE without coma, and subtle SE
Additional features of the seizure | between 01.01.2005 and 31.12.2023
  length, level of consciousness at onset, previous epileptic seizures
ICU Scoring Systems | between 01.01.2005 and 31.12.2023
  Critical illness severity scores (e.g., acute physiology and chronic health Evaluation (APACHE II), simplified acute physiology score (SAPS II), sequential organ failure assessment (SOFA), etc.)
Clinical neurologic monitoring scores | between 01.01.2005 and 31.12.2023
  Clinical neurologic monitoring scores (e.g., Richmond Agitation-Sedation Scale (RASS) , Seda-tion-Agitation Scale (SAS), Glasgow Coma Score (GCS), Intensive Care Delirium Screening Checklist (ICDSC), Status Epilepticus Severity Score (STESS))
Laboratory parameters | between 01.01.2005 and 31.12.2023
  C-Reactive Protein (CRP), albumin, Lactate Dehydrogenase (LDH), Creatin-Kinase (CK), procalcitonin, white blood cell levels, creatinine, liver enzymes, blood gas analyses, metabolic data
Outcome measure | between 01.01.2005 and 31.12.2023
  in-hospital death, survival, survival with neurofunctional alteration, Glasgow Outcome Score, return to neurofunctional premorbid baseline, readmission
Therapeutic features | between 01.01.2005 and 31.12.2023
  duration, dosage and number of treatment medication, number of antiseizure drugs, invasive procedures, such as intubation, mechanical, ventilation, vasopressors, installation of central lines, nutrition
Monitoring of vital signs | between 01.01.2005 and 31.12.2023
  blood pressure, heart rate, respiratory rate, oxygen saturation of the blood, body temperature, level of consciousness

CONTACTS AND LOCATIONS:
Overall Officials: Raoul Sutter, PD Dr. med, Principal Investigator — Clinic for Intensive Care Medicine, University Hospital Basel
Locations (2):
- Switzerland (2):
  - Cantonal Hospital Aarau (KSA), Aarau
  - Clinic for Intensive Care Medicine, University Hospital Basel, Basel